CLINICAL TRIAL: NCT03871127
Title: Ten-Year Outcomes of PREmier of Randomized Comparison of Sirolimus-Eluting Stent Implantation Versus Coronary Artery Bypass Surgery for Unprotected Left Main Coronary Artery Stenosis: PRE-COMBAT Trial
Brief Title: Ten-Year Outcomes of PRE-COMBAT Trial
Acronym: PRECOMBAT
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2019-02
Record Dates: First submitted 2019-03-07; First posted 2019-03-12 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease
Keywords: PCI; CABG; Left main
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Left main coronary disease
  Interventions: Procedure: Percutaneous coronary intervention; Procedure: coronary artery bypass graft

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Using sirolimus eluting stent
Procedure: coronary artery bypass graft — coronary artery bypass graft

SUMMARY:
This study evaluates Ten-Year Outcomes of PREmier of Randomized Comparison of Sirolimus-Eluting Stent Implantation Versus Coronary Artery Bypass Surgery for Unprotected Left Main Coronary Artery Stenosis(PRECOMBAT trial).

DETAILED DESCRIPTION:
This study is an extended one of PRECOMBAT trial.

ELIGIBILITY:
Inclusion Criteria:

* Subject group enrolled in PRECOMBAT trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject group enrolled in PRECOMBAT trial
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Composite outcome | 10 year
  The composite of death, myocardial infarction, and revascularization. Patients who have experienced any one of the following events are considered to have experienced the composite outcome: death, myocardial infarction, and revascularization

SECONDARY OUTCOMES:
All-cause mortality | 10 year
Cardiac death | 10 year
Myocardial infarction | 10 year
Cerebrovascular accident | 10 year
Target vessel revascularization | 10 year
Target lesion revascularization | 10 year
Stent thrombosis | 10 year
Binary restenosis in both in-stent and in-segment | 10 year
Graft reocclusion rate | 10 year
Graft patency rate | 10 year

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang Y, Jeong YJ, Hyun J, Lee J, Kim JH, Kim S, Kang DY, Lee PH, Ahn JM, Park DW, Park SJ; PRECOMBAT Investigators. Prognostic Value of Sex After Revascularization for Left Main Coronary Disease: Extended PRECOMBAT Study. JACC Asia. 2021 Nov 9;2(1):19-29. doi: 10.1016/j.jacasi.2021.08.009. eCollection 2022 Feb. PMID 36340254
- [Derived] Jeong YJ, Ahn JM, Hyun J, Lee J, Kim JH, Yang Y, Choe K, Park H, Kang DY, Lee PH, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Park SJ, Park DW. Ten-year Outcomes After Drug-Eluting Stents or Bypass Surgery for Left Main Coronary Disease in Patients With and Without Diabetes Mellitus: The PRECOMBAT Extended Follow-Up Study. J Am Heart Assoc. 2021 Jul 20;10(14):e019834. doi: 10.1161/JAHA.120.019834. Epub 2021 Jul 9. PMID 34238026
- [Derived] Lee J, Ahn JM, Kim JH, Jeong YJ, Hyun J, Yang Y, Lee JS, Park H, Kang DY, Lee PH, Park DW, Park SJ; on the behalf of the PRECOMBAT Investigators. Prognostic Effect of the SYNTAX Score on 10-Year Outcomes After Left Main Coronary Artery Revascularization in a Randomized Population: Insights From the Extended PRECOMBAT Trial. J Am Heart Assoc. 2021 Jul 20;10(14):e020359. doi: 10.1161/JAHA.120.020359. Epub 2021 Jul 6. PMID 34227392
- [Derived] Park DW, Ahn JM, Park H, Yun SC, Kang DY, Lee PH, Kim YH, Lim DS, Rha SW, Park GM, Gwon HC, Kim HS, Chae IH, Jang Y, Jeong MH, Tahk SJ, Seung KB, Park SJ; PRECOMBAT Investigators. Ten-Year Outcomes After Drug-Eluting Stents Versus Coronary Artery Bypass Grafting for Left Main Coronary Disease: Extended Follow-Up of the PRECOMBAT Trial. Circulation. 2020 May 5;141(18):1437-1446. doi: 10.1161/CIRCULATIONAHA.120.046039. Epub 2020 Mar 30. PMID 32223567